CLINICAL TRIAL: NCT04824898
Title: The Use of Injectable Plasma Rich Fibrin (I-PRF) Versus Simvastatin Gel in Surgical Management of Infra-bony Defects (A Randomized Controlled Clinical Trial)
Brief Title: The Use of Injectable Plasma Versus the Use of Simvastatin Gel in Surgical Management of Bony Defect in Dentistry
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMD-2019-1
Record Dates: First submitted 2021-03-17; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Intra-bony Pockets
Keywords: intra-bony pocket; I-prf; infra-bony pocket defect; vertical bone loss treatment; simvastation in pockets
MeSH Terms: interventions — Simvastatin; proliferation regulatory factors, human urine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- simvastatin 1.2%gel (Experimental): simvastatin 1.2%gel applied after open flap debridment in group I
  Interventions: Drug: Simvastatin
- I-prf (Experimental): Injectable plasma rich fibrin will be collected from each patient in group II and the applied after open flap debridment
  Interventions: Other: injectable plasma rich fibrin

INTERVENTIONS:
Drug: Simvastatin — Statins are first known as drugs that decrease the cholesterol level by inhibiting hydroxy-methyl-glutaryl co-enzyme-A reductase as they improve the lipid profile and help in the treatment of many cardiac diseases and has a role in osteoblasts diffrentiation
  Arms: simvastatin 1.2%gel
Other: injectable plasma rich fibrin — I- PRF is obtained by taking a blood sample from patients and then is centrifuged for three minutes at 3300 rpm, the I-PRF first will be in the form of liquid and then coagulate after few minutes from the injection
  Other Names: i-prf
  Arms: I-prf

SUMMARY:
Simvastatin (SMV) is one of the family members of statins, it has been showed in many previous studies that the simvastatin when dissolved with methylcellulose in situ gel with a concentration of 1.2% (SMV) approximately, can have a significant decrease in the pocket depth, regain the clinical attachment loss (CAL), and improve the bone level.

and the platelets concentrate has been introduced which is the injectable plasma rich fibrin (I-PRF), as it contains platelets and leukocytes, stem cells and endothelial cells that why it is called "blood concentrate ". So, it is proposed as treatment option in different periodontal procedures such as treatment of intra-bony defects,

DETAILED DESCRIPTION:
Group I ( Experimental group): will include 12 patients undergoing open flap debridement (OFD) followed by single application of I-PRF. Oral Hygiene measure will be instructed following treatment and maintenance visits will be given to them.

Group II (Control group): will include 12 patients undergoing open flap debridement (OFD) followed by application of 1.2% simvastatin gel. Oral Hygiene measure will be instructed following treatment and maintenance visits will be given to them.

* Oral hygiene instructions will be given to all patients.
* Full mouth Scaling and root planing (SRP) will be performed under local anesthesia.
* 4 to 8 weeks after the non-surgical periodontal therapy patients will be reassessed clinically and radiographically For all patients who are suitable for the study the following clinical and radiographic evaluation parameters will be measured: (All parameters will be recorded Pre-operatively (base line) and 6 months Post operatively by an examiner who will be masked to the type of treatment received by the individuals).

ELIGIBILITY:
Inclusion Criteria:

* • Age range between 25 and 40 years

  * Patients with severe chronic periodontitis having probing depth (PD) ≥6 mm and clinical attachment loss (CAL) ≥5 mm , or Stage III periodontitis
  * Patient having vertical bone loss ≥3 mm (distance between alveolar crest and base of the defect as confirmed by preoperative intraoral periapical radiographs using standardized parallel technique.)
  * Good compliance with the plaque control instructions following initial therapy
  * Availability for follow up and maintenance program.

Exclusion Criteria:

* • Patient with any systemic disease or conditions

  * Patient using antibiotic, anti-inflammatory, and immunosuppressive therapy during the preceding 3 months before the start of trial and during the study.
  * Patients who have undergone any periodontal treatment in the last 6 months
  * Pregnant and Lactating.
  * Reported allergy to any type of statins
  * Subjects who were tobacco or alcohol users
  * Vulnerable group of patients (e.g.: prisoners , handicapped , or decisionally impaired individuals )

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Plaque index (PI) | change from basline at 6 months
  clinical score
Gingival index (GI) | change from basline at 6 months
  clinical score
Probing depth (PD) | change from basline at 6 months
  clinical score
Clinical attachment level (CAL) | change from basline at 6 months
  clinical score

SECONDARY OUTCOMES:
radiographIc | from baseline at 6 months
  assess the alveolar bone level radiographically

CONTACTS AND LOCATIONS:
Overall Officials: suzan seif allah, professor, Study Director — faculty of dentistry ainshams university; ola m ezzat, ass professor, Study Chair — faculty of dentistry ainshams university
Locations (1):
- Ain Shams University, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code